CLINICAL TRIAL: NCT02861651
Title: Molecular Characterization of Acute Erythroid Leukemia (M6-AML) Using Targeted Next-generation Sequencing
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: M6-AML-14-004
Record Dates: First submitted 2016-07-08; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sequence Analysis, DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: DNA sequencing

SUMMARY:
Acute erythroid leukemia (AEL) is a morphologically distinct, infrequent (o5%) acute myeloid leukemia (AML) designed as M6 in the French- American-British (FAB) classification. The World Health Organization classification recognizes two subclasses, M6a, a leukemia with myeloid blast cells, and M6b, a very rare, purely erythroid AML. It may be difficult to distinguish between a myelodysplastic syndrome and AEL because of the erythroblastic proliferation, which is increased when dysplasia is present. No recurrent cytogenetic abnormality is specific of AEL and the prognosis is poor with a median survival of 17 months. A study of 14 genes in a series of 92 cases has shown that mutations are frequent in AEL and somewhat differ from the other AMLs by the lower and higher proportion of FLT3-ITD and TP53 mutations, respectively. Only three cases of AEL are reported in the TCGA database. To further characterize AEL, determine whether it constitutes a distinct class of AML and document the reasons for its poor prognosis, the investigators will search for molecular alterations in 40 M6a-AMLs using array comparative genomic hybridization (aCGH) and next-generation sequencing (NGS) of 106 genes known or suspected to have a role in myeloid malignancies or in erythrocyte differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 year
* Diagnosis of AML6
* Written consent obtained

Exclusion Criteria:

* No written consent
* No frozen samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AML-6 treated at Institut Paoli-Calmettes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Molecular characterization of AML-6 by NGS and CGH array | 1 year
  Molecular characterization using array comparative genomic hybridization (aCGH) and next-generation sequencing (NGS) of 106 genes known or suspected to have a role in myeloid malignancies or in erythrocyte differentiation.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Gelsi-Boyer, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du Rhône, France